CLINICAL TRIAL: NCT04440982
Title: Feasibility Study to Evaluate Performance of the LUM Imaging System for Intraoperative Detection of Residual Tumor in Breast Cancer Patients Receiving and Not Receiving Neoadjuvant Therapy
Brief Title: Feasibility Study of Intraoperative Detection of Residual Cancer in Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Required resources unavailable.
Sponsor: Lumicell, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CLP0008; 1R01CA212138-01 (NIH)
Record Dates: First submitted 2020-06-12; First posted 2020-06-22 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Neoadjuvant Therapy
Keywords: breast cancer surgery; lumpectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive the device intervention. All subjects will receive the study drug.
Who Masked: Investigator
Masking Description: Masking will only be applied until main lumpectomy is removed. At time of randomization, the study arm will be revealed to the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device Intervention: LUM Imaging System used during surgery (Experimental): The LUM Imaging Device will be used to look inside the lumpectomy cavity to see if the dye indicates any areas that may contain residual tumor. If the imaging identifies that there may be cancer cells remaining in the lumpectomy cavity, the surgeon will remove an additional piece of tissue. This process will be continued until a negative reading from the device is obtained or a maximum of 2 shaves of additional tissue has been removed. Patients in this arm will receive the study drug, LUM015
  Interventions: Drug: LUM015; Device: Lum Imaging System
- Standard of Care Arm (Other): The LUM Imaging Device will not be used to guide additional tissue removal. Patients in this arm will receive the study drug, LUM015.
  Interventions: Drug: LUM015

INTERVENTIONS:
Drug: LUM015 — LUM015 will be administered 2 to 6 hours prior to surgery for both arms. The LUM Imaging device will be used to assist in the removal of additional tumor tissue in the device intervention arm.
Device: Lum Imaging System — UM015 will be administered 2 to 6 hours prior to surgery for both arms. The LUM Imaging device will be used to assist in the removal of additional tumor tissue in the device intervention arm.
  Arms: Device Intervention: LUM Imaging System used during surgery

SUMMARY:
This is a prospective, multi-center, randomized, clinical trial evaluating patients undergoing breast conserving surgery using the LUM Imaging System.

DETAILED DESCRIPTION:
Detailed Description:

All subjects will be injected with LUM015. The injection of the study drug will occur 2-6 hours prior to surgery at a dose of 1.0 mg/kg. For all subjects, surgeons will perform main specimen resection per standard of care. For subjects randomized to the intervention arm, the surgeon will use the Lum System to scan and image all orientations within the cavity and The LUM Imaging System will guide shave removal. Then, for all subjects (control and intervention arm), comprehensive shaved margins are removed.

In this study, the initial cohort is a "training set" with 10 patients receiving neoadjuvant therapy to refine the tumor detection algorithm, if needed. After completion of enrollment of the initial 10 subjects for algorithm training, the Investigators will then enroll a cohort of patients who received neoadjuvant therapy to further evaluate the performance of the LUM Imaging System in this important subset of breast cancer patients. Concurrently to the enrollment of this cohort, surgeons will also enroll a cohort of patients who did not receive neoadjuvant therapy prior to surgery. Patients will be randomized 3:1 to a LUM-assisted lumpectomy versus a standard lumpectomy. In both arms, shaved margins will be taken from the entire lumpectomy cavity to compare the extent of residual tumor after standard and LUM-assisted lumpectomies to evaluate the negative predictive value of the LUM Imaging System following neoadjuvant therapy. Only the group of patients randomized to the device (intervention) arm will have the LUM Imaging System guide the removal of tissue prior to the removal of final comprehensive shaves of the entire cavity.

Study treatment ends when the surgery is completed. Patients are followed for adverse events until their standard of care follow-up visit or after any secondary surgery, whichever is longer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed primary invasive breast cancer, ductal carcinoma in situ (DCIS) or primary invasive breast cancer with a DCIS component.
* Female, age of 18 years or older.
* Subjects must have received neoadjuvant therapy for this breast cancer diagnosis prior to their lumpectomy procedure (cohorts 1 and 2).
* Subjects must be scheduled for a lumpectomy for a breast malignancy.
* Subjects must be able and willing to follow study procedures and instructions.
* Subjects must have received and signed an informed consent form.
* Subjects must have no uncontrolled serious medical problems except for the diagnosis of cancer, as per the exclusion criteria listed below.

  * Leukocytes > 1,000/mcL
  * Platelets > 50,000/mcL
  * total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * eGFR >= 60mL/min/1.73m2
* Subjects with ECOG performance status of 0 or 1.

Exclusion Criteria:

* Subjects who have been diagnosed with bilateral breast cancer and are undergoing bilateral resection procedure.
* Subjects who are pregnant at the time of diagnosis of their breast cancer. Breastfeeding should be discontinued if the mother is treated with LUM015.
* Subjects who are sexually active and not willing/able to use medically acceptable forms of contraception (hormonal or barrier method of birth control, abstinence) upon entering the study and for 60 days after injection of LUM015.
* Subjects who have taken an investigational drug within 14 days of enrollment.
* Subjects who will have administration of methylene blue or any blue or green dye for sentinel lymph node mapping on the day of the surgery prior to imaging the lumpectomy cavity with the LUM Imaging Device.
* Subjects who have not recovered from adverse events due to other pharmaceutical or diagnostic agents.
* Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 110 mm Hg; those subjects with known HTN should be stable within these ranges while under pharmaceutical therapy.
* Subjects with a history of allergic reaction to polyethylene glycol (PEG).
* Subjects with a history of allergic reaction to any oral or intravenous contrast agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with LUM015.
* Any subject for whom the investigator feels participation is not in the best interest of the subject.
* Subjects undergoing a second lumpectomy procedure because of positive margins in a previous surgery prior to entering this study.
* Subjects with prior ipsilateral breast cancer surgeries, mastectomies, breast reconstructions or implants.
* Subjects who have undergone a surgical biopsy for any reason in the ipsilateral breast performed less than 2 years prior to enrollment of this study.
* Subjects with prior ipsilateral reduction mammoplasties (breast reductions) performed less than 2 years prior to enrollment to this study.
* Subjects undergoing breast conserving surgery whose resected specimen (main lump, shaves, or any other resected tissue) will be evaluated with frozen section after the Lumicell-guided removal of shaves.
* Subjects with a history of allergic reaction to Tegaderm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Development and validation of tumor detection algorithms in breast cancer patients receiving neoadjuvant therapy | 1 month
  Refining of the previously validated tumor detection algorithm in breast cancer patients receiving neoadjuvant therapy will be conducted in the first cohort and the validation of this algorithm will use data from the second cohort.
Number of patients with reported adverse events | 14 days
  Reported adverse events will be assessed and aggregated according to event type, relation to device or drug, and severity.
Reduction in residual tumor | 3 months
  Evaluate reduction in residual tumor left after Lumicell assisted lumpectomy compared with SoC removal of main lumpectomy specimen in patients who have received and not received neo-adjuvant therapy
Report on patient reported outcomes and patient preference information | 12 months
  Collect and summarize patient reported information on outcomes and preference

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Smith, MD, PhD, Principal Investigator — Massachusetts General Hospital; Jorge Ferrer, PhD, Study Director — Lumicell, Inc.
Locations (6):
- United States (6):
  - Stanford Hospital and Clinics, Palo Alto, California
  - Morton Plant Mease Health Care Oncology Research, Clearwater, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke Cancer Center, Durham, North Carolina
  - Novant Health Cancer Center, Winston-Salem, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No